# An Observational Study to Determine Experience Patterns in Participants of Lung Cancer Clinical Trials

An Informed Consent Form For Power Clinical Trial's
Observational Medical Trial Participants

Date: February 25, 2023

#### Introduction

You are being asked to take part in a study to examine the experiences of people enrolled in clinical trials for lung cancer. You should be aware of the purpose and details of the research before deciding whether or not to take part. Please read this form completely, and feel free to ask any questions you may have. You have the choice of participating or not, and you are free to leave the research at any point without incurring any fees.

# Purpose of the Study:

This study aims to identify trends in individuals with lung cancer's clinical trial experiences.

The goal of this clinical trial is to learn more about the many factors that affect a patient's ability and interest to participate in and complete a medical research study during the clinical trial enrollment process. The goal of the experiment is to collect anonymized data from medical research in order to detect patterns in patient experiences that lead to a reduction in enrollment or completion rates.

If you choose to participate in this observational medical study, your therapy will not be altered or changed during the trial. Being a patient and taking part in medical research are two different things. This study's major objective is to gather information, analyze it, and learn more about the factors that influence a patient's capacity to participate.

#### Procedures of the Study:

Surveys will be given to you twice a week if you choose to participate. Each survey can be completed in up to thirty minutes. As long as you continue to take part in a different research study for lung cancer, we will additionally call you every three months. There are no interventions or therapies used in the study. You must ask your care team or doctor any queries you may have regarding your ongoing therapy.

#### Potential Risks:

There are no known health hazards from taking part in this study. Yet, since data is the only thing that can be used to conduct this research, confidentiality violation in clinical studies is a possible risk. While we handle enormous amounts of data, there is minimal possibility that this observational research will expose sensitive information.

#### Benefits:

You will not directly gain anything by taking part in this study. Your involvement could, however, progress this field of science.

# Confidentiality:

To the degree permitted by law, information about your involvement in this study will remain private. Your identity won't appear in any study data publications or presentations.

## Voluntary Involvement

You are not forced to take part in this study. You are also not subject to any consequences if you decide not to take part in the research or withdraw from it.

### Other Information About Lung Cancer Studies

Another kind of study for patients with lung cancer is a clinical trial including an intervention. Because a treatment plan is interventional in nature, the patient must adhere to it. The fact that this medical study is completely observational makes it distinctive. It won't suggest a different therapy for you or alter your current one.

Our staff is unaware of every clinical trial for lung cancer. But if you want to learn more about research on this illness, feel free to browse <u>lung cancer clinical trials</u> on Power's website or seek up <u>lung cancer studies</u> on clinicaltrials.gov.

# Other Research on Clinical Trial Participation

Here are some of the publications on participation rates that are available online if want to read up more:

<u>Unger, Joseph M., Elise Cook, Eric Tai, and Archie Bleyer. "The role of clinical trial participation in cancer research: barriers, evidence, and strategies." *American Society of Clinical Oncology Educational Book* 36 (2016): 185-198.</u>

Bleyer, Archie, Michael Montello, Troy Budd, and Scott Saxman. "National survival trends of young adults with sarcoma: lack of progress is associated with lack of clinical trial participation." *Cancer* 103, no. 9 (2005): 1891-1897.

# Participant Consent Statement

I acknowledge that I have been given the opportunity to read and understand this Informed Consent Form, and I have had the chance to ask any questions that I may

have. By signing below, I confirm that I voluntarily agree to participate in this clinical trial.

I understand that participation in this observational medical study is entirely voluntary, and I have the right to withdraw my consent at any time without prejudice. I understand that my treatment regime will not be modified or determined during this trial and that joining the medical study is separate from being a patient. I am aware that any personal information that I provide during the study will be kept confidential and that my anonymity will be protected.

I understand the nature of the study, the potential risks and benefits, and the procedures involved. I acknowledge that I have been given the opportunity to ask questions, and I feel sufficiently informed to make a decision about participating. By signing below, I agree to participate voluntarily in this study, and I give my consent for my anonymous medical study outcomes to be collected and analyzed for research purposes.

Participant Name:

| Participant Signature: |
|---|
| Date: |
| Person Taking Consent: |
| I have had a discussion with the participant regarding the information presented in this consent form. Based on our conversation, I believe that he or she has a clear understanding of the benefits, risks, alternatives, and procedures involved in this observational medical study. |
| Name: |
| Signature: |
| Date: |